CLINICAL TRIAL: NCT03350750
Title: A Placebo-Controlled Effectiveness in INPH Shunting (PENS) Trial: Proof of Concept
Brief Title: A Placebo-Controlled Effectiveness in INPH Shunting (PENS) Trial
Acronym: PENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Utah (Other); Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00083576
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Results first posted 2022-05-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus (INPH)

STUDY DESIGN:
Intervention Model Description: The primary intervention will be the initiation of the randomized initial shunt valve opening pressure setting to create a delayed treatment group in half of the study patients.
  Randomization will be to active or placebo (closed) shunt settings. At the time of the standard four-month evaluation, all subjects will be similarly non-invasively adjusted to bring all subjects in both groups to the active setting while maintaining blinding of the subjects. All settings will be verified by the adjusting neurosurgeon.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Open Shunt Group (Active Comparator): FDA-approved Certas Plus with Siphonguard, programmable CSF shunt valve setting to active (open shunt group)(setting 4)(110 mm H2O) at time of shunt implantation
  Interventions: Device: programmable CSF shunt valve
- Closed Shunt Group (Sham Comparator): FDA-approved Certas Plus with Siphonguard, programmable CSF shunt valve setting to placebo (closed shunt group)(setting 8)(>400 mm H2O) at time of shunt implantation followed by setting to active (setting 4) (110 mm H2O) four months after the procedure.
  Interventions: Device: programmable CSF shunt valve

INTERVENTIONS:
Device: programmable CSF shunt valve — Brain shunt surgery using a programmable CSF shunt valve
  Other Names: FDA-approved Certas Plus with Siphonguard

SUMMARY:
The Placebo-Controlled Effectiveness in Idiopathic Normal Pressure Hydrocephalus (iNPH) Shunting (PENS) trial is a multi-center blinded, randomized, placebo-controlled design investigation of cerebrospinal fluid (CSF) shunt surgery to study the shunt effectiveness in iNPH patients.

DETAILED DESCRIPTION:
The primary intervention will be setting the FDA-approved Certas Plus with Siphonguard, programmable CSF shunt valve to active (open shunt group)(setting 4)(110 mm H2O) or placebo (closed shunt group)(setting 8)(>400 mm H2O)in a 1:1 ratio. By the time of the primary objective evaluation at four months, the closed shunt group will have zero months of active treatment, and the open shunt group will have four months of active treatment. At four months, shunts for subjects in the closed shunt group will be adjusted to setting 4. To maintain blinding, all patients will be adjusted/ mock adjusted to the active setting in a similar fashion. Patients from both groups will not be adjusted before four months of active treatment, unless judged medically necessary by the treating team. Following four months of active treatment, all subjects in each group will have shunt adjustments according to clinical standards at each center.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years; and
* Diagnosis of INPH based on the Investigator's clinical judgement based on criteria and testing as described in the INPH Guidelines; and
* Evans Ratio ≥ 0.30; and
* One positive supplementary test to include large volume Lumbar Puncture or extended CSF drainage per institutional standards; and
* History or evidence of gait impairment (such as decreased step height or length,decreased speed, retropulsion as described in the INPH Guidelines) duration ≥ 6 months; and
* Participant has the sensory motor skills, communication skills and understanding to comply with the testing and reporting required in the PENS trial; and
* Participant is able to give written informed consent, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures.

Exclusion Criteria:

* Unable to walk 10 meters with or without an assistive device; or
* Baseline fastest gait velocity>1 m/sec and fastest gait velocity improvement is ≤ 30% with or without an assistive device; or
* Unable to return to the study center for follow up evaluation and shunt programming; or
* Participant is not medically cleared for shunt surgery per local standards; or
* Secondary NPH. (Prior encephalitis, meningitis, subarachnoid hemorrhage, traumatic brain injury (including concussion) within two years or with brain injury or skull fracture on baseline imaging, brain abscess, brain tumor, obstructive hydrocephalus (including acquired aqueductal stenosis and carcinomatous meningitis)); or
* Prior or existing shunts, endoscopic third ventriculostomy, or any previous surgical intervention for hydrocephalus; or
* Previous intracranial neurosurgical procedure; or
* Current treatment with anticoagulation medications or expected to be on anticoagulation medications in future based on clinician evaluation; or
* Symptomatic cerebral or cerebellar infarction within 6 months from screening(asymptomatic lacunar infarctions are permitted); or
* Diagnosis of Parkinsonian syndrome that, in the investigator's judgment, will complicate the outcome evaluation; or
* Diagnosis of schizophrenia or any psychiatric diagnosis (including depression) that in the investigator's judgment will complicate the outcome evaluation (such as neuroleptic treatment for schizophrenia); or
* Diagnosis of dementia disorder where the investigator considers cognition deficit limits participation in the study; or
* Conditions impairing gait that are considered to be unrelated to hydrocephalus, such as hemiparesis, spasticity, cerebellar ataxia or musculoskeletal and joint disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Luciano, MD, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (4):
  - Johns Hopkins Medicine, Baltimore, Maryland
  - University of New Mexico, Albuquerque, New Mexico
  - Cleveland Clinic, Cleveland, Ohio
  - University of Washington Medical Center, Seattle, Washington
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Vancouver General Hospital/University of British Colombia, Vancouver, British Colombia
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After subject enrollment and follow up have been completed, the Data Coordinating Center (DCC) of the study will prepare a final study database for analysis. A releasable database will be produced and completely de-identified in accordance with the definitions provided in the Health insurance Portability and Accountability Act (HIPAA). Namely, all identifiers specified in HIPAA will be re-coded in a manner that will make it impossible to deduce or impute the specific identity of any patient. The database will not contain any institutional identifiers.
  The DCC will also prepare a data dictionary that provides a concise definition of every data element included in the database. If specific data elements have idiosyncrasies that might affect interpretation or analysis, this will be discussed in the dictionary document.
  In accordance with policies determined by the investigators and funding sponsors, the releasable database will be provided to users in electronic form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after publication of the results of the primary analysis.
Access Criteria: individual participant data (IPD) will be made available to researchers submitting a request for data that includes an analytic plan approved by the Institutional Review Board (IRB) at their institution

REFERENCES:
- [Derived] Luciano M, Holubkov R, Williams MA, Malm J, Nagel S, Moghekar A, Eklund A, Zwimpfer T, Katzen H, Hanley DF, Hamilton MG; PENS Co-investigators and AHCRN Site PIs. Placebo-Controlled Effectiveness of Idiopathic Normal Pressure Hydrocephalus Shunting: A Randomized Pilot Trial. Neurosurgery. 2023 Mar 1;92(3):481-489. doi: 10.1227/neu.0000000000002225. Epub 2022 Nov 25. PMID 36700738

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Shunt Group: FDA-approved Certas Plus with Siphonguard, programmable cerebrospinal fluid (CSF) shunt valve setting to active (open shunt group)(setting 4)(110 mm H2O) at time of shunt implantation
  programmable CSF shunt valve: Brain shunt surgery using a programmable CSF shunt valve
Period: Overall Study
Arm/Group | Open Shunt Group | Closed Shunt Group
Started | 9 | 9
4-month Follow-up (Randomized Evaluation) | 8 | 8
12-Month Follow-up (Entire Study) | 8 | 8
Completed | 8 | 8
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Shunt Group | Closed Shunt Group | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74.0 [73.3 to 77.0] | 74.5 [70.1 to 76.5] | 74.2 [72.1 to 76.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 3 | 6
  Sweden | 1 | 1 | 2
  United States | 5 | 5 | 10
Evans' Ratio [Median (Inter-Quartile Range); unit: no unit] — Ratio (0-1) of the radiographic measure of the ventricular width of the largest frontal horn width (cm) and the greatest cerebral width in centimeters (cm) where a larger value indicates larger ventricular volume. The ratio has no unit.
  no unit | 0.36 [0.34 to 0.41] | 0.37 [0.35 to 0.42] | 0.37 [0.34 to 0.42]

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Velocity
Description: Evaluation of CSF shunting in Idiopathic Normal Pressure Hydrocephalus (INPH) patients through a group comparison of improvement from baseline at four months between active and placebo-controlled groups, using the primary endpoint of gait velocity in meters per second (m/s).
Time Frame: Baseline and 4 months
Population: Randomized patients alive at Month 4
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Open Shunt Group | Closed Shunt Group
Number analyzed (Participants) | 8 | 8
meters per second | 0.28 (0.284) | 0.04 (0.167)
Statistical Analysis 1: Comparison: Open Shunt Group vs Closed Shunt Group; Test type: Superiority; p = 0.071, ANCOVA; ANCOVA Model Effect (Open vs. Closed) = 0.22, 95% CI 2-sided [-0.02 to 0.46] — This is the coefficient for an indicator variable comparing the Open versus Closed shunt group, in a linear regression model with Month 4 gait velocity as the outcome and Baseline gait velocity included as a predictor along with treatment

2. Secondary Outcome: Change in Cognition as Assessed by the Montreal Cognitive Assessment (MoCA) Score
Description: Evaluate the effect of shunting between active and placebo-controlled groups at four months using MoCA test to assess cognition. Scores on the MoCA range from 0 to 30 where lower scores signify greater cognitive impairment.
Time Frame: Baseline and 4 Months
Population: Randomized patients alive at Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Shunt Group | Closed Shunt Group
Number analyzed (Participants) | 8 | 8
score on a scale | -0.13 (3.643) | 1.63 (1.598)
Statistical Analysis 1: Comparison: Open Shunt Group vs Closed Shunt Group; Test type: Superiority; p = 0.337, ANCOVA

3. Secondary Outcome: Change in Bladder Control as Assessed by the Overactive Bladder Questionnaire, Short Form
Description: Evaluate the effect of shunting between active and placebo-controlled groups at four months using Overactive Bladder Questionnaire, short form (OAB-q sf.) to assess bladder control. The OAB-q SF is scored from 0 to 100 with lower scores indicating worse QOL due to bladder control.
Time Frame: Baseline and 4 months
Population: Randomized patients alive at Month 4 with Outcome Data at Baseline and Month 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Shunt Group | Closed Shunt Group
Number analyzed (Participants) | 6 | 8
score on a scale | -23.3 (19.89) | 2.1 (17.81)
Statistical Analysis 1: Comparison: Open Shunt Group vs Closed Shunt Group; Test type: Superiority; p = 0.007, ANCOVA

4. Other Pre Specified Outcome: Change in Function as Assessed by the Lawton Activities of Daily Living/Independence in Activities of Daily Living (ADL/IADL) Test Score
Description: Evaluate the effect of shunting between active and placebo-controlled groups on change from baseline to four months using ADL/IADL test to assess function. Scores on the Lawton ADL/IADL scale range from 0 to 32 where a lower score indicates less independence in physical and instrumental daily living skills.
Time Frame: Baseline and 4 months
Population: Randomized Patients alive at Month 4 with Outcome Data for both Baseline and Month 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Shunt Group | Closed Shunt Group
Number analyzed (Participants) | 7 | 8
score on a scale | -5.7 (6.73) | 1.4 (3.89)
Statistical Analysis 1: Comparison: Open Shunt Group vs Closed Shunt Group; Test type: Superiority; p = 0.201, ANCOVA

5. Other Pre Specified Outcome: Change in Function as Assessed by the Modified Rankin Scale (MRS)
Description: Evaluate the effect of shunting between active and placebo-controlled groups at four months using MRS to assess function. Scores on the MRS range from 0 to 6 where higher scores signify increased disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
Time Frame: Baseline and 4 months
Population: Randomized Patients Alive at Month 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Shunt Group | Closed Shunt Group
Number analyzed (Participants) | 8 | 8
score on a scale | -0.88 (1.126) | -0.13 (0.641)
Statistical Analysis 1: Comparison: Open Shunt Group vs Closed Shunt Group; Test type: Superiority; p = 0.172, ANCOVA

6. Other Pre Specified Outcome: Change in Cognition as Assessed by the Symbol Digit Modalities Test (SDMT)
Description: Evaluate the effect of shunting between active and placebo-controlled groups at four months using SDMT to assess cognition. Scores on the SDMT range from 0 to 110 where lower scores are associated with reduced psychomotor speed.
Time Frame: Baseline and 4 months
Population: Randomized Patients Alive at Month 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Shunt Group | Closed Shunt Group
Number analyzed (Participants) | 8 | 8
score on a scale | -0.3 (6.61) | -0.1 (4.02)
Statistical Analysis 1: Comparison: Open Shunt Group vs Closed Shunt Group; Test type: Superiority; p = 0.780, ANCOVA

7. Other Pre Specified Outcome: Change in Gait Velocity From Shunt Activation to 8 Months After Active Shunting
Description: Evaluate the clinical improvement of all study participants at eight months of active shunting, using the primary outcome of gait velocity. For patients assigned to Open shunt, active shunting is from Baseline to Month 8 of the study. For patients assigned to Closed Shunt, active shunting is from Month 4 of the study (immediately prior to opening of initially Closed shunt) to Month 12 (i.e., after 8 months of the patient having an open shunt).
Time Frame: Up to 8 months after active shunting
Population: All randomized patients alive with gait velocity evaluated 8 months after active shunting.
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- All Randomized Patients: All patients in the trial (arms combined for this evaluation). All randomized patients evaluated after 8 months of active shunting
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 13
meters per second | 0.38 (0.229)
Statistical Analysis 1: Comparison: All Randomized Patients; Test type: Superiority; p < 0.001, t-test, 2 sided

8. Other Pre Specified Outcome: Change in Cognition Using MoCA From Baseline to 8 Months After Active Shunting
Description: Evaluate the clinical improvement of all study participants at eight months of active shunting using MoCA to assess cognition. Scores on the MoCA range from 0 to 30 where lower scores signify greater cognitive impairment.
Time Frame: Baseline and 8 months after active shunting
Population: all patients with MoCA available at baseline and after 8 months of active shunting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 13
score on a scale | 1.0 (2.92)
Statistical Analysis 1: Comparison: All Randomized Patients; Test type: Superiority; p = 0.240, t-test, 2 sided

9. Other Pre Specified Outcome: Change in Bladder Control From Baseline to 8 Months After Active Shunting
Description: Evaluate the clinical improvement of all study participants at eight months of active shunting using OAB-q test to assess bladder control. The OAB-q SF is scored from 0 to 100 with lower scores indicating worse QOL due to bladder control.
Time Frame: Baseline and 8 months after active shunting
Population: Patients with outcome data available at baseline and at 8 months after active shunting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 12
score on a scale | -25.0 (29.42)
Statistical Analysis 1: Comparison: All Randomized Patients; Test type: Superiority; p = 0.013, t-test, 2 sided

10. Other Pre Specified Outcome: Change in Function Using ADL/IADL From Baseline to 8 Months After Active Shunting
Description: as for outcome 4
Time Frame: Baseline and 8 months after active shunting
Population: All participants with outcome data available at baseline and after 8 months of active shunting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 12
score on a scale | -4.7 (5.88)
Statistical Analysis 1: Comparison: All Randomized Patients; Test type: Superiority; p = 0.019, t-test, 2 sided

11. Other Pre Specified Outcome: Change in Function Using MRS From Baseline to 8 Months After Active Shunting
Description: as for outcome 5
Time Frame: Baseline and 8 months after active shunting
Population: All randomizred patients with MRS data at baseline and at 8 months of active shunting.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 13
score on a scale | -0.6 (0.96)
Statistical Analysis 1: Comparison: All Randomized Patients; Test type: Superiority; p = 0.040, t-test, 2 sided

12. Other Pre Specified Outcome: Change in Cognition Using SDMT From Baseline to 8 Months After Active Shunting
Description: Evaluate the clinical improvement of all study participants at eight months of active shunting using SDMT to assess cognition. Scores on the SDMT range from 0 to 110 where lower scores are associated with reduced psychomotor speed.
Time Frame: Baseline and 8 months after active shunting
Population: All patients with SDMT data available at baseline and 8 months after active shunting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 13
score on a scale | 5.8 (7.21)
Statistical Analysis 1: Comparison: All Randomized Patients; Test type: Superiority; p = 0.013, t-test, 2 sided

13. Other Pre Specified Outcome: Number of Patients With Falls
Description: Evaluate the effect of shunting between active and placebo-controlled groups at four months by assessing the number of patients with falls.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Shunt Group | Closed Shunt Group
Number analyzed (Participants) | 9 | 9
Participants | 0 | 2
Statistical Analysis 1: Comparison: Open Shunt Group vs Closed Shunt Group; Test type: Superiority; p = 0.235, Fisher Exact; Fisher's exact test with a mid-p-value correction

14. Other Pre Specified Outcome: Frequency of Adverse Effects
Description: Evaluate the clinical improvement of all study participants at eight months of active shunting by assessing the frequency of falls, surgical and non-surgical complications, related and unrelated.
Time Frame: 8 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Adverse Events
Description: Compare adverse events (AEs) in the active versus placebo-controlled group at four months and at eight months of active shunting.
Time Frame: 4 and 8 months of active shunting
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From time of randomization until 1 year after initial shunting procedure.
Description: There are two intervention groups in the study. Open shunt arm starts with shunt "active" at the time of shunt insertion. Closed shunt arm begins with an initial 4-month period where shunt is set to placebo and then to active after 4 months of shunt insertion. Adverse events were assessed for these two arms. Adverse events occurring during the period of the closed shunt were not separately monitored from adverse events occurring during the period of the open shunt for the Closed shunt group.
Arm/Group | Open Shunt Group | Closed Shunt Group
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/9
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/9
Other Adverse Events (participants affected / at risk) | 6/9 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Shunt Group (N=9) | Closed Shunt Group (N=9)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hospitalization for Grade 3 Generalized Muscle Weakness
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) — Stroke
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) — Hospitalization for Septic urinary tract infection (UTI)
Subdural Effusion (Nervous system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gallbladder necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Shunt Group (N=9) | Closed Shunt Group (N=9)
Transient Decrease in MOCA Score (Investigations) | 4 (6) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — External head trauma
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — Abdominal cramping
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) — Residual balance issues
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) — Fever of unknown origin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03350750/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT03350750/SAP_002.pdf
  • Informed Consent Form (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03350750/ICF_003.pdf